CLINICAL TRIAL: NCT01028469
Title: Artelon MTP Spacer - Surgical Treatment of Mild to Moderate Hallux Rigidus
Brief Title: Artelon Metatarsophalangeal (MTP) Spacer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artimplant AB (Industry)
Responsible Party: Katrin Gisselfalt, Chief Research & Development, Artimplant
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP026
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Osteoarthritis; Hallux Rigidus
MeSH Terms: conditions — Osteoarthritis; Hallux Rigidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artelon MTP Spacer (Experimental): Metatarsophalageal hemi-implant
  Interventions: Device: Artelon MTP Spacer

INTERVENTIONS:
Device: Artelon MTP Spacer — Metatarsophalangeal hemi-implant

SUMMARY:
The aim of this prospective, case series is to evaluate the surgical treatment of painful and disabling osteoarthrosis in the MTP-I joint by insertion of an Artelon MTP Spacer.

ELIGIBILITY:
Inclusion Criteria:

* The patient experiences pain and limitations of the great toe dorsiflexion at the MTP-I joint.
* The patient has a clinically and radiographically verified arthritis in the MTP-I joint indicating the need for surgical treatment.
* The patient reads, understands and is able to complete the study questionnaires in Swedish.
* The patient has received written and oral information regarding the study and has signed the informed consent form.

Exclusion criteria:

* The patient has a pronounced hallux rigidus without mobility in the MTP-I joint (ROM = 0°).
* The patient has previously received surgical treatment affecting the anatomy of the MTP-I joint.
* The patient has a systemic rheumatic disease, ongoing infection, hallux valgus or is seriously ill.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Pain, function and alignment of the treated toe evaluated by the investigator using the American Orthopeadic Foot & Ankle Society (AOFAS) clinical rating system. | pre-treatment and 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Martin Alund, M.D., Principal Investigator — Sahlgrenska University Hospital, Mölndal, Sweden
Locations (1):
- Sahlgrenska Universitetssjukhuset, Område Ortopedi, Mölndal, Mölndal, Sweden